CLINICAL TRIAL: NCT02405689
Title: The Effect of Sevoflurane-dexmedetomidine and Sevoflurane-remifentanil on Biochemical Markers During Open Heart Surgery
Brief Title: Myocardial Protection and Anesthetic Agents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, mediha turktan, assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: open heart surgery
Record Dates: First submitted 2015-03-18; First posted 2015-04-01 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-03

CONDITIONS: Myocardial Ischemic Reperfusion Injury
MeSH Terms: conditions — Myocardial Reperfusion Injury | interventions — Remifentanil; Dexmedetomidine; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- remifentanil (Active Comparator): In the remifentanil group, anesthesia was maintained with 0.5-1.5% sevoflurane and 0.125-0.25 μg/kg/min remifentanil infusion during surgery
  Interventions: Drug: Remifentanil; Drug: Sevoflurane
- dexmedetomidine (Active Comparator): In the dexmedetomidine group anesthesia was maintained with 0.5-1.5% sevoflurane and 0.5 μg/kg dexmedetomidine loading dose during 10 minute and then 0.3-0.9 μg/kg/min infusion.
  Interventions: Drug: Dexmedetomidine; Drug: Sevoflurane

INTERVENTIONS:
Drug: Remifentanil
  Arms: remifentanil
Drug: Dexmedetomidine
  Arms: dexmedetomidine
Drug: Sevoflurane

SUMMARY:
The aim of this study was to investigate the myocardial protective effects of remifentanil and dexmedetomidine in cardiac surgery.

DETAILED DESCRIPTION:
Fifty patients is included in this study. Routine monitorization included a 5-lead electrocardiogram (ECG), invasive arterial monitoring, pulse oximetry, capnography, temperature monitoring. Invasive arterial catheter were inserted under local anesthesia. Central venous catheter (jugular or subclavian) and esophageal heat probe were inserted after tracheal intubation.

Anesthesia induction was standardized in all patients and included 1 mg/kg propofol, 1 μg/kg fentanyl and 0.1 mg/kg vecuronium bromus to facilitate endotracheal intubation. The patients were divided into two groups by computer randomization method. Group R (n=25), remifentanil group and Group D (n=25) dexmedetomidine group. In the remifentanil group, anesthesia was maintained with 0.5-1.5% sevoflurane and 0.125-0.25 μg/kg/min remifentanil infusion. In the dexmedetomidine group anesthesia was maintained with 0.5-1.5% sevoflurane and 0.5 μg/kg dexmedetomidine loading dose during 10 minute and 0.3-0.9 μg/kg/min infusion.

Cardiopulmonary bypass (CPB) period was started after aort and venous cannulae were inserted. Mean arterial pressure, central venous pressure, venous oxygen saturation (SVO2) and arterial blood gase analysis were recorded. All blood samples include laktat, pyruvate, CKMB and Troponin-T were taken via the coronary sinus catheter at specific time intervals (precardiopulmonary bypass, 20 minutes after cross clamp, 20 minutes after removal cross clamp and 10 minutes after cardiopulmonary bypass).

Cardiopulmonary bypass time, aortic cross clamping time, the need of defibrillation/intraaortic balloon pumping (IABP)/extracorporeal membrane oxygenator (ECMO), urine output, positive inotropic agents requirement were recorded. At the end of surgery, the patients were transferred intensive care unit intubated and full monitorized.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to open heart surgery
* American Society of Anesthesiologists (ASA) physical status of II-III

Exclusion Criteria:

* Emergency surgery, prior cardiac surgery, ejection fraction < 50%, restrictive or obstructive pulmonary disease, preoperative mechanical ventilation, intra-aortic balloon pump, chronic liver and renal failure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
level of laktat | at 20 minutes after cross clamp, 20 minutes after removal cross clamp and 10 minutes after cardiopulmonary bypass
Level of pyruvate | at 20 minutes after cross clamp, 20 minutes after removal cross clamp and 10 minutes after cardiopulmonary bypass
level of CKMB | at 20 minutes after cross clamp, 20 minutes after removal cross clamp, 10 minutes after cardiopulmonary bypass
level of Troponin-T | at 20 minutes after cross clamp, 20 minutes after removal cross clamp, 10 minutes after cardiopulmonary bypass

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

REFERENCES:
- [Background] Kapoor P, Mandal B, Chowdhury U, Singh S, Kiran U. Changes in myocardial lactate, pyruvate and lactate-pyruvate ratio during cardiopulmonary bypass for elective adult cardiac surgery: Early indicator of morbidity. J Anaesthesiol Clin Pharmacol. 2011 Apr;27(2):225-32. doi: 10.4103/0970-9185.81819. PMID 21772685
- [Background] Triggiani M, Simeone F, Gallorini C, Paolini G, Donatelli F, Paolillo G, Dolci A, Grossi A. Measurement of cardiac troponin T and myosin to detect perioperative myocardial damage during coronary surgery. Cardiovasc Surg. 1994 Aug;2(4):441-5. PMID 7953444